CLINICAL TRIAL: NCT04428619
Title: Neuromodulation With Percutaneous Electrical Nerve Field Stimulation for Adults With Irritable Bowel Syndrome: A Randomized, Double-Blind, Sham-Controlled Pilot Study
Brief Title: Percutaneous Electrical Nerve Field Stimulation for Adults With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Innovative Health Solutions (Industry)
Responsible Party: Principal Investigator, Lin Chang, MD, Vice-Chief, Vatche and Tamar Manoukian Division of Digestive Diseases, Program Director, UCLA GI Fellowship Program, Co-Director, G. Oppenheimer Center for Neurobiology of Stress and Resilience, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 19-001796
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain; Autonomic Nervous System Imbalance
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients who meet study eligibility criteria will be randomly assigned (1:1) in blocks of two and four, using a code generated by a randomization program to 4 weeks of stimulation with an active or inactive (sham) PENFS device. Per manufacturer design, both active stimulation and sham are below a detectable sensation threshold. Allocation will be concealed, and all physicians, statisticians, participants, and research coordinators will be unaware of device codes. One research coordinator who has no patient contact will be unblinded and handle allocation and storage of devices. At the end of 4 weeks, patients will be asked to which device arm they believe they were randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Peripheral Electrical Nerve Field Stimulation (PENFS) Device (Active Comparator): The PENFS device has a battery activated generator and wire harness. Four leads are attached to the generator, each with a sterile 2 mm, titanium needle. The patient's ear is trans-illuminated to identify neurovascular bundles that are avoided during needle placement. The generator is attached with adhesive to the skin behind the patient's ear. Needles are inserted into the dorsal and ventral aspects of the ear, within 1-1.5 mm of the vascular branches to create a field effect. The device settings are standardized and deliver 3.2 volts with alternating frequencies (1 ms pulses of 1 Hz and 10 Hz) every 2 s. This stimulation targets central pain pathways through branches of cranial nerves V, VII, IX, and X, which innervate the external ear. The device is worn for 5 days/week for a total of 4 weeks. Patients remove devices at home on day 6 of each treatment cycle. Patients will be asked to wear a SmartWatch during the study to monitor heart rate.
  Interventions: Device: Peripheral Electrical Nerve Field Stimulation (PENFS) Device
- Sham Device (Sham Comparator): The sham devices will be identical to the active devices but will not administer electrical charges. Per manufacturer design and patient anecdotal experience from previous studies, both active stimulation and sham are below detectable sensation threshold. Per report from previous studies, some patients may experience a sensation around the ear after percutaneous needle placement; however, this sensation can occur with equal likelihood in the active or sham device. The device is worn for 5 days a week for a total of 4 weeks. Patients remove devices at home on day 6 of each treatment cycle. Patients will also be asked to wear a SmartWatch as above.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Peripheral Electrical Nerve Field Stimulation (PENFS) Device — Patients will complete daily worst abdominal pain and bowel habit questionnaires for 1 week prior to initial PENFS device placement to provide a baseline. At visit 1, patients will complete the Bowel Symptom Questionnaire, IBS Symptom Severity Scale (IBS-SSS), PROMIS Belly Pain Scale, Gas and Bloating, Constipation, and Diarrhea Scales, Hospital Anxiety and Depression Scale, and Visceral Sensitivity Index, heart rate variability will be measured, and they will have the initial PENFS device placed. Patients will complete daily worst abdominal pain (scale 0-10) questionnaires throughout the duration of the study. They will return every 7 days for a total of 4 visits for device replacement and additional questionnaires, including the IBS-SSS. Four devices will be placed in total (start of weeks 1, 2, 3, and 4). Stimulation time is 5 days/week during each of the 4 consecutive weeks. Additional questionnaires will be completed at the end of week 4 and at extended follow-up (8 weeks).
  Arms: Peripheral Electrical Nerve Field Stimulation (PENFS) Device
Device: Sham Device — Patients will complete daily worst abdominal pain and bowel habit questionnaires for 1 week prior to initial sham device placement to provide a baseline. At visit 1, patients will complete the Bowel Symptom Questionnaire, IBS Symptom Severity Scale (IBS-SSS), PROMIS Belly Pain Scale, Gas and Bloating, Constipation, and Diarrhea Scales, Hospital Anxiety and Depression Scale, and Visceral Sensitivity Index, heart rate variability will be measured, and they will have the initial sham device placed. Patients will complete daily worst abdominal pain (scale 0-10) questionnaires throughout the duration of the study. They will return every 7 days for a total of 4 visits for device replacement and additional questionnaires, including the IBS-SSS. Four devices will be placed in total (start of weeks 1, 2, 3, and 4). Stimulation time is 5 days/week during each of the 4 consecutive weeks. Additional questionnaires will be completed at the end of week 4 and at extended follow-up (8 weeks).
  Arms: Sham Device

SUMMARY:
This is a prospective, double-blind, randomized, sham-controlled pilot study evaluating the efficacy of percutaneous electrical nerve field stimulation for the treatment of adult patients with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
IBS has a worldwide prevalence around 11% and is characterized by chronic or recurrent abdominal pain associated with altered bowel habits. Abnormalities within the brain-gut axis, visceral hypersensitivity, and dysfunction of the autonomic nervous system are important components contributing to the pathophysiology of IBS. Despite recent advances in medical therapies for IBS, a significant subgroup of patients fails to experience satisfactory relief of abdominal pain. Given evidence of anti-inflammatory and anti-nociceptive components of vagal nerve pathways, peripheral field stimulation of the vagus nerve may help reduce abdominal pain in patients with IBS.

Percutaneous electrical nerve field stimulation (PENFS) administered via the IB-Stim device (Innovative Health Solutions, Versailles, IN, USA) has been shown to be efficacious in adolescent patients with abdominal-pain-related functional GI disorders, including IBS. This device uses discontinuous frequencies of stimulation to target central pain pathways through branches of cranial nerves V, VII, IX, and X that innervate the external ear and project to certain brainstem nuclei, including the nucleus tractus solitarius (NTS). The NTS then acts as a relay station to other brain areas involved in pain modulation and autonomic control, including the rostral ventral medulla, locus coeruleus, hypothalamus, and amygdala. In adolescent studies, PENFS was associated with a greater reduction in worst abdominal pain and composite abdominal pain scores from baseline as well as compared with a sham device after three weeks of treatment. These effects were sustained over an extended follow-up period with minimal to no side effects. In addition, a greater proportion of adolescents in the PENFS arm achieved at least a 30% reduction in worst abdominal pain scores from baseline after 3 weeks of treatment.

The IB-Stim is the first device to be approved by the Food and Drug Administration (FDA) for the treatment of functional abdominal pain in adolescents aged 11-18 with IBS. However, the efficacy of PENFS in adults with IBS is not currently known. This study is a double-blind, randomized, sham-controlled pilot study evaluating the efficacy of PENFS using IB-Stim for the treatment of IBS symptoms in adult patients with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18-60 years, who are able to provide written, informed consent.
* Patients must meet Rome IV criteria for IBS, confirmed by a gastroenterologist who specializes in functional GI disorders. Any of the IBS bowel habit subtypes (diarrhea, constipation, mixed bowel habits, unclassified) will be allowed.
* Average daily worst abdominal pain score between 4 and 8 (on a 0-10-point rating scale).
* Minimum of 2 days of abdominal pain/week prior to starting trial.
* At least moderate IBS symptom severity with an IBS-SSS of at least 175 (total score range 0-500).
* If receiving pharmacologic therapy for abdominal pain associated with IBS, doses must be stable for at least 60 days prior to enrollment in the trial.
* If receiving pharmacologic therapy for IBS that does not have an effect on abdominal pain, doses must be stable for at least 30 days prior to enrollment in the trial.

Mandatory Exclusion Criteria:

* Patients under the age of 18 years or over the age of 60 years
* Patients who cannot provide informed consent or do not speak English
* Co-morbid, organic medical conditions associated with abdominal pain, including: Inflammatory bowel disease, chronic liver disease, peptic ulcer disease, celiac disease, diverticulitis, appendicitis, colorectal cancer, endometriosis, pregnancy, other intestinal or extra-intestinal malignancies. Patients with overlapping functional GI disorders (i.e. functional dyspepsia) will not be excluded as long as IBS is their predominant disorder
* History of surgery involving CN V, VII, IX, or X.
* History of abdominal surgeries other than appendectomy or cholecystectomy at least 6 months before entry into trial.
* Patients on chronic opioids, benzodiazepines, or with illicit substance use
* Patients with underlying neurologic conditions, including history of: seizures, CVA, uncontrolled migraines, traumatic brain injury, multiple sclerosis
* Patients with underlying psychiatric conditions
* Patients with dermatologic conditions affecting the ear, face, or neck region (i.e. psoriasis), or with cuts or abrasions to the external ear that would interfere with needle placement
* Patients with hemophilia or other bleeding disorders
* Patients with any implanted electrical device
* Patients who are pregnant or breastfeeding

Preferred, but not mandatory, exclusion criteria:

* Movement disorder
* Unwillingness to wear the SmartWatch on upper extremity (left or right wrist)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chang, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Krasaelap A, Sood MR, Li BUK, Unteutsch R, Yan K, Nugent M, Simpson P, Kovacic K. Efficacy of Auricular Neurostimulation in Adolescents With Irritable Bowel Syndrome in a Randomized, Double-Blind Trial. Clin Gastroenterol Hepatol. 2020 Aug;18(9):1987-1994.e2. doi: 10.1016/j.cgh.2019.10.012. Epub 2019 Oct 14. PMID 31622740

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Started | 7 | 8
Completed | 6 | 6
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Peripheral Electrical Nerve Field Stimulation (PENFS) Device: The PENFS device has a battery activated generator and wire harness. Four leads are attached to the generator, each with a sterile 2 mm, titanium needle. The patient's ear is trans-illuminated to identify neurovascular bundles that are avoided during needle placement. The generator is attached with adhesive to the skin behind the patient's ear. Needles are inserted into the dorsal and ventral aspects of the ear, within 1-1.5 mm of the vascular branches to create a field effect. The device settings are standardized and deliver 3.2 volts with alternating frequencies (1 ms pulses of 1 Hz and 10 Hz) every 2 s.
- Total: Total of all reporting groups
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 6 | 9
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in IBS Symptom Severity From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in IBS symptom severity in adult IBS patients after 4 weeks of treatment and at extended follow-up (8 weeks), assessed through a mean change in the IBS-SSS between groups. Answers were measured using the IBS-SSS. Higher scores indicate worse symptoms. The score range is 0-500.
Time Frame: 4 weeks, 8 weeks.
Population: 7 with device, 8 with sham.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device: The PENFS device has a battery activated generator and wire harness. Four leads are attached to the generator, each with a sterile 2 mm, titanium needle. The patient's ear is trans-illuminated to identify neurovascular bundles that are avoided during needle placement. The generator is attached with adhesive to the skin behind the patient's ear. Needles are inserted into the dorsal and ventral aspects of the ear, within 1-1.5 mm of the vascular branches to create a field effect. The device settings are standardized and deliver 3.2 volts with alternating frequencies (1 ms pulses of 1 Hz and 10 Hz) every 2 s. This stimulation targets central pain pathways through branches of cranial nerves V, VII, IX, and X, which innervate the external ear. The device is worn for 5 days/week for a total of 4 weeks
  The sham devices will be identical to the active devices but will not administer electrical charges. Per manufacturer design and patient anecdotal experience from previous studies, both active stimulation and sham are below detectable sensation threshold. Per report from previous studies, some patients may experience a sensation around the ear after percutaneous needle placement; however, this sensation can occur with equal likelihood in the active or sham device. The device is worn for 5 days a week for a total of 4 weeks. Patients remove devices at home on day 6 of each treatment cycle. Patients will also be asked to wear a SmartWatch as above.
- Sham Device: The sham devices will be identical to the active devices but will not administer electrical charges. Per manufacturer design and patient anecdotal experience from previous studies, both active stimulation and sham are below detectable sensation threshold.
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  4 weeks | 280 (39.9) | 320 (91.7)
  8 weeks | 244 (122) | 316 (76.5)

2. Secondary Outcome: Mean and Standard Deviation of Heart Rate Variability (HRV) Measures in PENFS Device and Sham Groups at 4 Weeks.
Description: Same measures as outcome measure 12. LF peak FFT: Peak frequency within the low-frequency range (typically 0.04-0.15 Hz) of the HRV spectrum HF peak FFT: Peak frequency within the high-frequency range (typically 0.15-0.4 Hz) of the HRV spectrum.
  VLF peak AR: Peak frequency within the very-low-frequency range (typically 0.0033-0.04 Hz) of the HRV spectrum.
  HF peak AR: Peak frequency within the high-frequency range of the HRV spectrum. LF peak AR: Peak frequency within the low-frequency range of the HRV spectrum.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Peripheral Electrical Nerve Field Stimulation (PENFS) Device: The PENFS device has a battery activated generator and wire harness. Four leads are attached to the generator, each with a sterile 2 mm, titanium needle. The patient's ear is trans-illuminated to identify neurovascular bundles that are avoided during needle placement. The generator is attached with adhesive to the skin behind the patient's ear. Needles are inserted into the dorsal and ventral aspects of the ear, within 1-1.5 mm of the vascular branches to create a field effect. The device settings are standardized and deliver 3.2 volts with alternating frequencies (1 ms pulses of 1 Hz and 10 Hz) every 2 s. This stimulation targets central pain pathways through branches of cranial nerves V, VII, IX, and X, which innervate the external ear. The device is worn for 5 days/week for a total of 4 weeks
  The sham devices will be identical to the active devices but will not administer electrical charges. Per manufacturer design and patient anecdotal experience from previous studies, both active stimulation and sham are below detectable sensation threshold. Per report from previous studies, some patients may experience a sensation around the ear after percutaneous needle placement; however, this sensation can occur with equal likelihood in the active or sham device. The device is worn for 5 days a week for a total of 4 weeks. Patients remove devices at home on day 6 of each treatment cycle. Patients will also be asked to wear a SmartWatch as above.
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 7 | 8
Hz
  LFpeak_FFT_Hz_ACT_Wk_4 | 0.0817 (0.0454) | 0.103 (0.0115)
  HFpeak_FFT_Hz_ACT_Wk_4 | 0.296 (0.0263) | 0.287 (0.0555)
  VLFpeak_AR_Hz_ACT_Wk_4 | 0.0400 (0) | 0.0278 (0.0212)
  LFpeak_AR_Hz_ACT_Wk_4 | 0.0975 (0.0357) | 0.0833 (0.0393)
  HFpeak_AR_Hz_ACT_Wk_4 | 0.298 (0.0357) | 0.294 (0.0483)

3. Secondary Outcome: IBS Symptom Severity Responder Rate
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in IBS symptom severity in adult IBS patients after 4 weeks of treatment compared to baseline. Participants will be considered responders if there is at least a 50-point reduction on the IBS-SSS.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 6 | 6
Participants | 3 | 2

4. Secondary Outcome: Mean Change in Average Daily Worst Abdominal Pain From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on mean worst daily abdominal pain scores after 4 weeks compared to baseline in adult patients with IBS. The scale is measured as follows, with higher scores indicating worse pain:
  Daily Worse Abdominal Pain Severity:
  • How would you rate your worst abdominal pain over the past 24-hours (0-10)?
  o 0 = no pain, 10= worst pain possible
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale | 5.02 (1.84) | 5.03 (1.61)

5. Secondary Outcome: Change in Average Daily Stool Consistency From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in average daily stool consistency after 4 weeks of treatment compared to baseline, assessed using the Bristol Stool Form Scale (BSFS) (stool types 1-7; types 1 and 2 indicate constipation, types 3 and 4 are normal consistency stools, type 5 indicates stool lacking fiber, types 6 and 7 indicate diarrhea).
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale | 2.91 (1.10) | 3.78 (2.39)

6. Secondary Outcome: Change in Average Weekly Bowel Habits From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in average weekly bowel habits after 4 weeks of treatment and at extended follow-up (8 weeks) compared to baseline, assessed through the PROMIS Gastrointestinal Constipation Scale (percentiles 0.3-100%; higher percentiles indicate greater constipation).
Time Frame: Week 4, week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  week 4 | 51.5 (9.11) | 62.8 (3.93)
  week 8 | 53.8 (6.43) | 61.3 (4.74)

7. Secondary Outcome: Change in Quality of Life From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in IBS-quality of life (IBS-QOL) in adult patients with IBS after 4 weeks of treatment and at extended follow-up (8 weeks) compared to baseline. IBS QOL will be assessed on a scale from 0-100, with higher scores indicating better IBS specific quality of life.
Time Frame: Week 4, week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  week 4 | 66.8 (20.4) | 42.1 (19.0)
  week 8 | 42.3 (22.7) | 74.7 (20.3)

8. Secondary Outcome: "Number of Participants With Treatment-related Adverse Events as Assessed by a Weekly Adverse Events Questionnaire
Description: To compare the incidence of treatment-related adverse events from PENFS therapy versus sham therapy in adult patients with IBS. Adverse events will be assessed by a weekly adverse events questionnaire that determines the severity of the adverse event, the relationship to the study intervention, the action taken regarding the study intervention, the outcome of the adverse event, whether or not the adverse event was expected, and if the event was considered a serious adverse event (SAE).
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

9. Secondary Outcome: Change in Average Weekly Bloating Symptoms From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in average weekly bloating symptoms at 4 weeks and at extended follow-up (8 weeks) compared to baseline, assessed through the PROMIS Gastrointestinal Gas and Bloating Scale (percentiles 0.1-100%; higher percentiles indicate greater gas and bloating).
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  4 weeks | 58.2 (8.11) | 65.0 (6.44)
  8 weeks | 56.7 (8.56) | 64.2 (5.64)

10. Secondary Outcome: Change in Average Weekly Abdominal Pain Symptoms From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in average weekly abdominal pain symptoms at 4 weeks and at extended follow-up (8 weeks) compared to baseline, assessed through the PROMIS Gastrointestinal Belly Pain Scale (percentiles 2-100%; higher percentiles indicate worse abdominal pain).
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  4 weeks | 65.8 (4.72) | 69.4 (3.82)
  8 weeks | 62.8 (9.92) | 69.3 (2.53)

11. Secondary Outcome: Chang in Average Weekly Bowel Habits From Baseline
Description: To compare the efficacy of PENFS therapy versus sham therapy on the change in average weekly bowel habits after 4 weeks of treatment and at extended follow-up (8 weeks) compared to baseline, assessed through the PROMIS Gastrointestinal Diarrhea Scale (percentiles 1-100%; higher percentiles indicate greater diarrhea).
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device and Sham Device | Sham Device
Number analyzed (Participants) | 7 | 8
score on a scale
  4 weeks | 59.9 (8.15) | 63.4 (5.92)
  8 weeks | 50.8 (9.31) | 54.8 (14.0)

12. Secondary Outcome: Mean and Standard Deviation of Heart Rate Variability (HRV) Measures in PENFS Device and Sham Groups at Baseline.
Description: LF peak FFT: Peak frequency within the low-frequency range (typically 0.04-0.15 Hz) of the HRV spectrum, as determined by Fast Fourier Transform (FFT) analysis.
  HF peak FFT: Represents the peak frequency within the high-frequency range (typically 0.15-0.4 Hz) of the HRV spectrum, as determined by FFT analysis.
  VLF peak AR: Represents the peak frequency within the very-low-frequency range (typically 0.0033-0.04 Hz) of the HRV spectrum, as determined by autoregressive (AR) modeling.
  HF peak AR: Represents the peak frequency within the high-frequency range of the HRV spectrum, as determined by AR modeling.
  LF peak AR: Represents the peak frequency within the low-frequency range of the HRV spectrum, as det
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 7 | 8
Hz
  LFpeak_FFT_Hz_ACT_Ba | 0.0822 (0.0217) | 0.0913 (0.04)
  HFpeak_FFT_Hz_ACT_Ba | 0.219 (0.0489) | 0.197 (0.0258)
  VLFpeak_AR_Hz_ACT_Ba | 0.0400 (0) | 0.0253 (0.0201)
  LFpeak_AR_Hz_ACT_Ba | 0.119 (0.0345) | 0.0787 (0.0450)
  HFpeak_AR_Hz_ACT_Ba | 0.213 (0.0516) | 0.214 (0.0508)

13. Secondary Outcome: Mean and Standard Deviation of Heart Rate Variability (HRV) Measures in PENFS Device and Sham Groups at Baseline.
Description: HF/LF ratio FFT: Ratio of high-frequency to low-frequency ratio in heart rate variability (HRV) analysis, as determined by FFT analysis. It reflects the balance between parasympathetic (HF) and sympathetic (LF) nervous system activity influencing heart rate.
  HF/LF ratio ACT: Ratio of high-frequency to low-frequency ratio in heart rate variability (HRV) analysis, as determined by AR modeling. It reflects the balance between parasympathetic (HF) and sympathetic (LF) nervous system activity influencing heart rate.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 7 | 8
ratio
  LF_HF_ratio_FFT_ACT_Ba | 1.26 (2.30) | 6.66 (13.33)
  LF_HF_ratio_AR_ACT_Ba | 1.70 (3.09) | 5.13 (9.86)

14. Secondary Outcome: Mean and Standard Deviation of Heart Rate Variability (HRV) Measures in PENFS Device and Sham Groups at 4 Weeks.
Description: HF/LF ratio AR: Ratio of high-frequency to low-frequency ratio in heart rate variability (HRV) analysis, as determined by AR. It reflects the balance between parasympathetic (HF) and sympathetic (LF) nervous system activity influencing heart rate.
  HF/LF ratio FFT: Ratio of high-frequency to low-frequency ratio in heart rate variability (HRV) analysis; reflects the balance between parasympathetic (HF) and sympathetic (LF) nervous system activity influencing heart rate.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
Number analyzed (Participants) | 7 | 8
ratio
  LF_HF_ratio_FFT_ACT_Wk_4 | 2.83 (4.32) | 0.574 (0.0332)
  LF_HF_ratio_AR_ACT_Wk_4 | 2.21 (3.18) | 0.592 (0.128)

ADVERSE EVENTS:
Time Frame: Each participant was assessed over 8 weeks (baseline - week 8).
Arm/Group | Peripheral Electrical Nerve Field Stimulation (PENFS) Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT04428619/Prot_SAP_000.pdf